CLINICAL TRIAL: NCT05019989
Title: DIANA-5: Randomized Trial to Test the Efficacy of Dietary Change and Physical Activity to Prevent or Delay the Development of Recurrences in Breast Cancer Patients Estimated to be at High Risk of Recurrence Hormonal and Metabolic Reasons
Brief Title: Trial of Diet, Physical Activity and Breast Cancer Recurrences: the DIANA-5 Study
Acronym: DIANA-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); European Institute of Oncology (Other); Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other); Federico II University (Other); IRCCS Cancer Referral Center of Basilicata (Other); ARNAS Civico Di Cristina Benfratelli Hospital (Other); Lega Italiana per la Lotta contro i Tumori (Other); Azienda Socio Sanitaria Territoriale di Mantova (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Anna Villarini, Biologist, Nutritionist, PhD and Senior researcher, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT 37/07
Record Dates: First submitted 2021-07-14; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer Invasive
Keywords: Breast cancer; Diet; Physical activity; Recurrences
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Recurrence | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Trial of Diet, Physical Activity and Breast Cancer Recurrences. The investigators recruited 1542 patients' high risk and randomized them in two groups: 773 (control group) have received general standard written recommendation for healthy lifestyle without, however, any active support; 769 (intervention group) have received a combination of individual and group contacts over the course of one year, including kitchen courses, gym and dance classes, common meals and reinforcing meetings, with emphasis on a comprehensive dietary and life-style change.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: on diet and physical activity (Experimental): Individual advice on diet and on physical activity Kitchen courses to teach basic Mediterranean and macrobiotic recipes (two 1-day course plus ten 3-h courses associated with common dinner) (15-20 participants at a time) Fortnightly common lunch or dinner (50-60 participant at a time) Basic gymnastic course (twelve - monthly- 2-hour courses)
  * Study newsletter, with scientific information, kitchen recipes, study facilities
  * Periodic conferences on diet and health
  * Periodic reinforcement meetings with common meals, gymnastic sessions, and dancing, after the first year
  * Periodic body weight assessment (weekly self-measurement and monthly measurement at the study center)
  * Discounted rate for advanced kitchen courses
  * Psychological support groups
  Interventions: Behavioral: Intervention group on diet and physical activity
- Control group: only public recommendations on lifestyle (Experimental): 1. Invitation leaflet, explaining the rationale of the study and including basic life-style recommendations, based on the 1997 World Cancer Research Fund recommendations (to be updated in 2007) and the Italian National Institute of Nutrition food pyramid.
  2. Dissemination of the information on the study by media
  3. Yearly follow-up questionnaire on breast events and dietary and physical activity chang
  Interventions: Behavioral: Control group: only public recommendation an lifestyle

INTERVENTIONS:
Behavioral: Intervention group on diet and physical activity — The intervention wanted to increase physical activity, controlling weight, promoting healthy diet.
  1. Physical activity: achieve and maintain regular participation in a moderate intensity physical activity program of 210 minutes/week (30 min on average per day) over at least 3 days /week; decrease sedentary behaviors by 30 minutes/day on at least 5 days/week
  2. Weight control: reducing energy intake relative to expenditure is the primary dietary focus for promoting weight loss in overweight or obese participants, and maintaining a healthy energy balance is the primary focus for normal weight participants. Participants will be encouraged to include whole grains and high-fiber vegetables
  3. Healthy diet: reducing calorie intake, through the preferred consumptions of unrefined cereals, pulses and vegetables, reducing high glycemic index food and high insulinemic foods, such as sugar and milk; reducing sources of saturated fat and animal protein (except fish)
  Arms: Intervention group: on diet and physical activity
Behavioral: Control group: only public recommendation an lifestyle — 1. Invitation leaflet, explaining the rationale of the study and including basic life-style recommendations, based on the 1997 World Cancer Research Fund recommendations (to be updated in 2007) and the Italian National Institute of Nutrition food pyramid.
  2. Dissemination of the information on the study by media
  3. Yearly follow-up questionnaire on breast events and dietary and physical activity chang
  Arms: Control group: only public recommendations on lifestyle

SUMMARY:
The investigators recruited 1542 Breast Cancer (BC) patients and to randomize the participants in two groups: 773 have received standard recommendations for healthy lifestyle without, however, any active support; 700 have received a combination of individual and group contacts over the course of one year, including kitchen courses, gym and dance classes, common meals and reinforcing meetings, with emphasis on a comprehensive dietary change including low saturated fat and low refined carbohydrates, and high whole grain cereals and pulses consumption. Compliance have been monitored through weight change and plasma glucose, triglycerides, cholesterol and testosterone.

The main analysis will be by intention to treat. Under the hypothesis of reducing recurrence rate by 25% or 33% the statistical power of the study is 80% or, respectively, 90%, (P<0.05, 5-year follow-up).

DETAILED DESCRIPTION:
Aims The investigators have been proposing a randomized intervention trial of diet and physical activity to reduce BC relapse (local, distant), and second ipsilateral or contralateral BC risk, in BC patients at high metabolic-endocrine of recurrence risk.

Secondary aims:

* to evaluate the effect of the combined dietary and physical activity change on the prevalence of Metabolic Syndrome
* to evaluate the effect of the combined dietary and physical activity change on the prevalence on risk biomarkers (BMI > 24.9 kg/m^2)
* to evaluate the effect of the combined dietary and physical activity change on the prevalence on risk biomarkers (testosterone >= 0.4 ng/ml)
* to evaluate the effect of the combined dietary and physical activity change on the prevalence on risk biomarkers (insulin > pmol/l)
* to evaluate the effect of the intervention on the development of other life-style related health conditions (other cancers, diabetes, hypertension, dyslipidemia, total mortality)

Recruitment:

Potential participants have been recruited at the time of diagnosis through follow-up clinics, patients' associations, or the media. Patients have been requested to sign an informed consent, including authorization for getting blood samples, for storing samples for future studies. The investigators collected demographic information, fasting measure body weight, height, waist circumference, and blood pressure, blood glucose, LDL and HDL cholesterol, triglycerides, testosterone and insulin. Eligible patients have filled in a baseline questionnaire on medical history, medication use, reproductive and body weight history, usual physical activity, and a validated semi-quantitative food frequency questionnaire.

Biological bank: the investigators collected and stored at -80°C one aliquot of whole blood, three 2-ml serum aliquot and two 2-ml buffy coat aliquot.

Randomization:

The investigators recruited 1542 patients' high risk and randomized the participants in two groups: 773 (control group) have received general standard written recommendation for healthy lifestyle without, however, any active support; 770 (intervention group) have received a combination of individual and group contacts over the course of one year, including kitchen courses, gym and dance classes, common meals and reinforcing meetings, with emphasis on a comprehensive dietary and life-style change.

Randomization has been carried out within strata of age, treatment (no adjuvant therapy, chemotherapy only, hormonal therapy only, both hormonal and chemotherapy) and axillary nodal status at diagnosis.

Patients who did not satisfy the high-risk criteria have been given the same general recommendations as the control group, and have been followed up as an external low risk group.

Intervention:

The intervention wanted aim to increase physical activity, controlling weight, and promoting healthy diet.

1. Physical activity: achieve and maintain regular participation in a moderate intensity physical activity program of 210 minutes/week (30 min on average per day) over at least 3 days /week; decrease sedentary behaviors by 30 minutes/day on at least 5 days/week. During the first 12 months one group physical activity session per month offered to enhance program adoption. Women who wanted to take up vigorous sports encouraged to do so. For those who do not progressed to more vigorous activity, the focus was on maintaining moderate activities, such as walking. For self-monitoring and compliance enhancement, study participants had use logs, fill-in questionnaires and armband to monitor physical activity.
2. Weight control: reducing energy intake relative to expenditure was the primary dietary focus for promoting weight loss in overweight or obese participants, while maintaining a healthy energy balance was the primary focus for normal weight participants. Participants were encouraged to include whole grains, pulses and high-fiber vegetables.
3. Healthy diet: reducing calorie intake, through the preferred consumptions of highly satiating foods, such as unrefined cereals, legumes and vegetables, reducing high glycemic index food, high insulinemic foods, saturated fat, preferring instead unrefined vegetable fats, such as extra virgin olive oil, nuts and oleaginous seeds, reducing protein intake, mainly animal protein (except fish).

Baseline and yearly measurements:

Height and weight: electronic scale with women in light clothes and without shoes. In a sample of cases body fat and lean mass will be measured with bioelectric impedance (BIA).

Blood pressure: electronic device. Serum glucose, triglycerides and cholesterol: standard quality-controlled laboratory techniques.

Serum Testosterone and Insulin: Radioimmunoassay (RIA). For testosterone the investigators have used a direct RIA kit which has been validated by comparison with indirect assay after organic extraction of serum samples and celite purification.

Compliance:

Compliance has been monitored through lifestyle questionnaires, dietary questionnaires, weight change and plasma glucose, triglycerides, cholesterol, insulin, testosterone changes after one year of intervention. A compliance score has been computed, based on the direction of change in all these biomarkers.

Follow-up and outcome events:

The main outcome is the new BC events including:

* new primary breast cancer
* local/regional recurrence
* distant/metastatic recurrence The follow up have been based on the routine clinical follow-up at the collaborating hospitals, the periodic questionnaires to study participants, the regional cancer registry and hospital discharge diagnosis system, and death certificates.

Statistical power:

The survival of BC patients in Italy is dramatically increasing: 5-year relative survival increased from 80.6% for patients diagnosed in the early 1990s to 85.6% for patients diagnosed in the early 2000s. For these patients the estimated relapse free survival is 81.9. Such a survival improvement is accompanied by a postponement of the incidence of relapse.

The original aim was to recruit 1,200 high risk patients in order to have 600 patients per arm, which shall guarantee 80% chance of getting a significant difference also with 25% reduction, and allowing for 90% compliance in the intervention group and 10% contamination of the control group.

Statistical analysis:

Nowadays the investigators are assessing the baseline association between androgens, insulin, and several measures of adiposity including body mass index (BMI), waist circumference and percentage body fat, through Spearman correlation coefficients. Furthermore, the investigators are comparing the change in food consumption, body weight, and geometric means of hormones end points from baseline to 12 months in the intervention and control group.

The main analysis of the intervention effect on the incidence of recurrences is by intention to treat, i.e. based on assigned treatment at the time of randomization, regardless of adherence. Later, as a secondary analysis the investigators shall assess the effect by change in body weight and biomarkers. The investigators shall compute total survival and disease-free survival.

Hazard ratios and confidence intervals will be computed by the Cox proportional hazard model, with standard clinic-pathological prognostic covariates as potential confounders. Separate analyses will be carried out by Estrogen Receptors, Progesterone Receptors and erbB2 status. The investigators decided to carry out another follow-up in 2022 as the relapse time has lengthened to 10 years, due to new therapies, and to evaluate the effects on lifestyle due to closures during the pandemia severe acute respiratory syndrome-CoV-2.

Feasibility:

The principal investigator (at first dr. Franco Berrino and later dr. Anna Villarini) has long term experience in carrying on and coordinating epidemiological studies, including small-scale dietary intervention studies. The Milano National Cancer Institute and the others collaborating center is fully equipped with facilities for kitchen courses and gym facilities.

Control of potential biases:

Performance bias-patients have been recruited after the main treatments have been planned or delivered. In no case the allocation to the intervention or control group or the compliance will affect treatment.

Measurement bias-patients and researchers cannot be blinded, but the ascertainment of outcome was carried out by clinicians that were not involved in the study.

Attrition bias-Based on previous studies the investigators expect a fairly high compliance in the intervention group (>90%) but also some modification in the control group. After the main analysis by intention to treat, therefore, secondary analyses will be carried out by compliance score.

ELIGIBILITY:
Inclusion Criteria:

* Mastectomy or conservative surgery for invasive breast cancer, any type, in the last five years (the investigators recruited mostly patients at the time or after surgery, when chemotherapy has been concluded and hormonal therapy, if necessary, has been started)
* Absence of signs or symptoms suggestive of recurrences
* Presence of one or more of the following endocrine/metabolic indicators: serum testosterone level ≥ 0.4 ng/ml (1 nmol/ml), corresponding to the median value in BC patients, or serum insulin ≥ 50 pmol/L, corresponding to the upper quartile of insulin distribution in Breast Cancer patients, or metabolic syndrome, present in about 15% of Breast Cancer patients.

Exclusion Criteria:

* Metastatic disease or previous relapse
* Age >70
* Physical or mental handicaps that would have impeded to engage in moderate physical activity or participate in kitchen classes

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women breast cancer diagnosis
Enrollment: 1542 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction of recurrences | Baseline, fifth year
  The investigators have been proposing a randomized intervention trial of diet and physical activity to change BC relapse (local, distant), and second ipsilateral or contralateral BC, in BC patients at high risk of recurrence because of biochemical markers of increased risk, namely high serum testosterone and/or high fasting insulin and/or metabolic syndrome. Several other markers of increased recurrence risk are available, such as cancer stage at diagnosis, histological grade, hormonal receptors and other gene expression profile. All these will be registered, but the investigators are specifically interested in markers of the host that can be modified through life-style.

SECONDARY OUTCOMES:
Modification lifestyle and Metabolic Syndrome (MetS) | Baseline, first year
  The effect of the combined dietary and physical activity change on the prevalence of MetS (defined as the presence of three or more risk factors: waist circumference >85 cm, systolic blood pressure >130 mmhg and /or diastolic blood pressure >85 mmhg), glycaemia >100mg/100ml, triglycerides >150 mg/100ml or HDL cholesterol <50 mg/100ml) that is hypothesized to be intermediate factor in the association of diet and physical activity with BC recurrences.
Modification lifestyle and Body Mass Index (BMI) | Baseline, first year
  The effect of the combined dietary and physical activity change on the prevalence on risk biomarkers (BMI > 24.9 kg/m^2) that is hypothesized to be intermediate factors in the association of diet and physical activity with BC recurrences.
Modification lifestyle and Testosterone | Baseline, first year
  The effect of the combined dietary and physical activity change on the prevalence on risk biomarkers (testosterone >= 0.4 ng/ml) that is hypothesized to be intermediate factors in the association of diet and physical activity with BC recurrences.
Modification lifestyle and Insulin | Baseline, first year
  The effect of the combined dietary and physical activity change on the prevalence on risk biomarkers (insulin > 50 pmol/L) that is hypothesized to be intermediate factors in the association of diet and physical activity with BC recurrences.
Development other cancer | Baseline, fifth year
  The effect of the intervention on the incidence of other cancers in all patients through the medical history reported in the medical record
Development diabetes | Baseline, fifth year
  The effect of the intervention on the incidence of diabetes in all patients through the medical history reported in the medical record
Total mortality | Baseline, fifth year
  The effect of the intervention on total mortality in all patients through the reference oncologists

CONTACTS AND LOCATIONS:
Overall Officials: ANNA VILLARINI, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, dataset, statistical analysis plan, informed consent form and clinical study report were discussed through meetings held with all the collaborating centers. The individual participant data (IPD) were delivered to the coordinators of the individual centers in coded anonymous.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be become available from baseline up to 10 years after study the end of recruitment (2027) for all coordinators of collaborating centers
Access Criteria: The data are available on the National Cancer Institute of MILANO (Foundation-Institute of Hospitalization and Scientific Care), network managed

REFERENCES:
- [Result] Roveda E, Bruno E, Galasso L, Mule A, Castelli L, Villarini A, Caumo A, Esposito F, Montaruli A, Pasanisi P. Rest-activity circadian rhythm in breast cancer survivors at 5 years after the primary diagnosis. Chronobiol Int. 2019 Aug;36(8):1156-1165. doi: 10.1080/07420528.2019.1621330. Epub 2019 Jun 10. PMID 31177874
- [Result] Roveda E, Vitale JA, Bruno E, Montaruli A, Pasanisi P, Villarini A, Gargano G, Galasso L, Berrino F, Caumo A, Carandente F. Protective Effect of Aerobic Physical Activity on Sleep Behavior in Breast Cancer Survivors. Integr Cancer Ther. 2017 Mar;16(1):21-31. doi: 10.1177/1534735416651719. Epub 2016 Jun 1. PMID 27252076
- [Result] Bruno E, Gargano G, Villarini A, Traina A, Johansson H, Mano MP, Santucci De Magistris M, Simeoni M, Consolaro E, Mercandino A, Barbero M, Galasso R, Bassi MC, Zarcone M, Zagallo E, Venturelli E, Bellegotti M, Berrino F, Pasanisi P. Adherence to WCRF/AICR cancer prevention recommendations and metabolic syndrome in breast cancer patients. Int J Cancer. 2016 Jan 1;138(1):237-44. doi: 10.1002/ijc.29689. Epub 2015 Jul 28. PMID 26175188
- [Result] Berrino F, Villarini A, Traina A, Bonanni B, Panico S, Mano MP, Mercandino A, Galasso R, Barbero M, Simeoni M, Bassi MC, Consolaro E, Johansson H, Zarcone M, Bruno E, Gargano G, Venturelli E, Pasanisi P. Metabolic syndrome and breast cancer prognosis. Breast Cancer Res Treat. 2014 Aug;147(1):159-65. doi: 10.1007/s10549-014-3076-6. Epub 2014 Aug 8. PMID 25104441
- [Result] Villarini A, Pasanisi P, Traina A, Mano MP, Bonanni B, Panico S, Scipioni C, Galasso R, Paduos A, Simeoni M, Bellotti E, Barbero M, Macellari G, Venturelli E, Raimondi M, Bruno E, Gargano G, Fornaciari G, Morelli D, Seregni E, Krogh V, Berrino F. Lifestyle and breast cancer recurrences: the DIANA-5 trial. Tumori. 2012 Jan-Feb;98(1):1-18. doi: 10.1177/030089161209800101. PMID 22495696
- [Derived] Djuric O, Bonvicini L, Pellegrini M, Bruno E, Pasanisi P, Gargano G, Curtosi P, Berrino F, Giorgi Rossi P, Villarini A. Diet, body composition and metabolic and hormonal profile in women at high risk of breast cancer recurrence: A secondary mediation analysis of the DIANA-5 trial. Clin Nutr. 2026 Jan;56:106537. doi: 10.1016/j.clnu.2025.11.021. Epub 2025 Dec 4. PMID 41483481
- [Derived] De Santi M, Annibalini G, Marano G, Biganzoli G, Venturelli E, Pellegrini M, Lucertini F, Brandi G, Biganzoli E, Barbieri E, Villarini A. Association between metabolic syndrome, insulin resistance, and IGF-1 in breast cancer survivors of DIANA-5 study. J Cancer Res Clin Oncol. 2023 Sep;149(11):8639-8648. doi: 10.1007/s00432-023-04755-6. Epub 2023 Apr 27. PMID 37106164

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT05019989/Prot_SAP_000.pdf